CLINICAL TRIAL: NCT01751516
Title: PET/MRI as a Predictor for Response to Preoperative Radiation Therapy and Chemotherapy in Resectable Rectal Cancer: a Pilot Study.
Brief Title: PET/MRI as a Predictor of Response to Pre-op Chemoradiation in Resectable Rectal Cancer: a Pilot Study
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1225
Record Dates: First submitted 2012-12-13; First posted 2012-12-18 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Rectal Carcinoma
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a single arm, single center pilot study of 40 patients with uT3N0 or uT1-3N+ rectal cancer receiving pre-operative chemoradiation. Subjects will undergo PET/MRI scans before and after surgery.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine the negative predictive value of PET/MRI for determining pathological complete response from neoadjuvant chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

* Low-lying, low- to moderate-risk pathologically-confirmed rectal cancer (stage uT3n) or uT1-3N+
* Negative workup for distant disease
* > 18 years of age
* Pre-treatment workup completed including:
* history and physical
* CT or MRI of the abdomen and pelvis
* endoscopic tumor evaluation (biopsy, blood work to assess CEA and hematopoietic, renal and liver function)
* if female of child-bearing age, negative pregnancy test
* Recommendation to undergo preoperative concurrent chemoradiation, as determined by the treating physician
* Informed consent reviewed and signed

Exclusion Criteria:

* Not deemed a candidate for preoperative chemoradiation for medical reasons, such as uncontrolled infection (including HIV), uncontrolled diabetes mellitus or cardiac disease
* Hemoglobin ≤ 10.0 g/dL (transfusion allowed to achieve or maintain levels)
* ANC ≤ 1,500/cubic mm³
* Platelet count ≤ 100,000/mm³
* ALT and AST ≥ 2.5 times upper level of normal (ULN)
* Alkaline phosphatase ≥ 2.5 times ULN
* Total bilirubin ≥ 1.5 times ULN
* Creatinine clearance < 50 mL/min
* Creatinine ≥ 1.5 times ULN
* Not deemed a candidate for concurrent preoperative chemoradiation for social reasons, such as psychiatric illness
* Not deemed a surgical candidate
* Currently active second malignancy, except non-melanoma skin cancer, non-invasive bladder cancer, low risk adenocarcinoma of the prostate and carcinoma in situ of the cervix
* Previous pelvic radiation therapy
* History of severe reaction to gadolinium
* Inability to tolerate MRI (e.g., inability to lie flat for > 1 hour)
* Presence of a pacemaker, intracranial aneurysm clip, bladder stimulator, cochlear implant or metal near eyes
* Body Mass Index (BMI) > 35
* Pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UNC Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2018-03-04 (Actual)

PRIMARY OUTCOMES:
Negative post-chemoradiation PET/MRI scan, as correlated with surgical pathology | 4-8 weeks post-chemoradiation

SECONDARY OUTCOMES:
Recurrence-free survival | 5 years
Disease-specific survival | 5 years
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joel E Tepper, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina-Chapel Hill, Chapel Hill, North Carolina, United States